CLINICAL TRIAL: NCT00885495
Title: The Effects of Darunavir Plus Ritonavir on the Pharmacokinetics and Pharmacodynamics of Rosuvastatin
Brief Title: Darunavir/Ritonavir and Rosuvastatin Pharmacokinetic Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Carl J. Fichtenbaum, Professor, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IDC 40
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Results first posted 2022-01-19 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: HIV Infections
Keywords: HIV; dyslipidemia; statins; protease inhibitors
MeSH Terms: conditions — HIV Infections; Dyslipidemias | interventions — Darunavir; Ritonavir; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Active Comparator): Darunavir+ritonavir x 7 days; Rosuvastatin x 7 days; Combination x 7 days
  Interventions: Drug: darunavir, ritonavir, rosuvastatin
- A (Active Comparator): Rosuvastatin x 7 days; darunavir+ritonavir x 7 days; Combination x 7 days
  Interventions: Drug: rosuvastatin, darunavir, ritonavir

INTERVENTIONS:
Drug: darunavir, ritonavir, rosuvastatin — darunavir 600 mg twice daily for 7 days ritonavir 100 mg twice daily for 7 days rosuvastatin 10 mg once daily for 7 days Combination of all three drugs for 7 days
  Other Names: Prezista; Norvir; Crestor
  Arms: B
Drug: rosuvastatin, darunavir, ritonavir — rosuvastatin 10 mg daily for 7 days; darunavir 600 mg twice daily for 7 days with ritonavir 100 mg twice daily for 7 days; Combination of all three for 7 days
  Other Names: Prezista; Norvir; Crestor
  Arms: A

SUMMARY:
This is a phase I, open-label, controlled drug interaction study to determine the effects of darunavir plus ritonavir on the pharmacokinetics of the hydroxymethylglutaryl coenzyme A (HMG-CoA) reductase inhibitor, rosuvastatin, in HIV-1-seronegative subjects.

DETAILED DESCRIPTION:
Twelve HIV-negative healthy volunteers will be randomized to one of two groups. Group 1 would receive rosuvastatin 10mg daily (Treatment A) in interval 1 for 7 days, followed by a washout period of at least 7 days. In interval 2, darunavir/ritonavir 600/100mg bid (Treatment B) would be administered for 7 days, followed by another 7 day washout period. Lastly, in interval 3 subjects will administer darunavir/ritonavir and rosuvastatin (Treatment C) for total of 7 days. Group 2 will administer Treatment B in interval 1 for 7 days, followed by a washout period of 7 days, then treatment A in interval 2 for 7 days followed by another 7 day washout period. Group 2 would then co-administer rosuvastatin and darunavir/ritonavir for the last 7 days. Intensive PK sampling will be performed on day 7, 21 and 35 following a meal.

ELIGIBILITY:
Inclusion Criteria:

1. Absence of HIV-1/HIV-2 infection as documented by a licensed ELISA test kit within 21 days prior to study entry.
2. Male or female subjects, aged ≥ 18 and ≤ 60 years
3. Weight ≥50 kg and a Body Mass Index ([BMI], weight in kg divided by the square of height in meters) ≥18.0 and ≤ 35.0 kg/m2. Refer to Appendix I.
4. Informed Consent Form (ICF) signed voluntarily before the first trial-related activity.
5. Able to comply with protocol requirements.
6. Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, vital signs, and the results of blood tests and a urinalysis carried out at screening.

Exclusion Criteria:

1. History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in the investigator's opinion would compromise subject's safety and/or compliance with the trial procedures.
2. Currently active significant gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease, that in the opinion of the investigator would represent a contraindication to study enrollment.
3. Creatinine clearance of ≤ 60mL/min.
4. Currently significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability.
5. eruptions, drug allergies, food allergy, dermatitis, eczema, psoriasis, or urticaria, that in the opinion of the investigator would represent a contraindication to study enrollment.
6. Previously demonstrated clinically significant allergy or hypersensitivity to any of the excipients of the medications administered in the trial.
7. History of significant drug allergy such as, but not limited to, sulphonamides and penicillins. Prezista is a sulphonamide. The potential for cross-sensitivity between drugs in the sulphonamide class and Prezista in HIV-negative subjects is unknown.
8. Use of concomitant medication, including investigational, prescription, and over-the-counter products and dietary supplements with the following exceptions: aspirin, acetaminophen, anti-histamines such as diphenhydramine, inhalers for asthma, daily multivitamins, mineral supplements and hormonal oral contraceptives. Concomitant medication other than those listed above must have been discontinued at least 7 days before study entry.
9. Female subjects of childbearing potential without use of effective nonhormonal birth control methods, or not willing to continue practicing these birth control methods for at least 30 days after the end of the treatment period; Note: Estrogen-based hormonal contraception may not be reliable when taking Prezista, therefore to be eligible for this trial, women of childbearing potential should either:

   * use a double barrier method to prevent pregnancy (i.e., using a condom with either diaphragm or cervical cap);
   * use non-estrogen hormonal based contraceptives in combination with a barrier contraceptive (i.e., male condom, diaphragm or cervical cap, or female condom);
   * use a intrauterine device in combination with a barrier contraceptive (i.e., male condom, diaphragm or cervical cap, or female condom);
   * be not sexually active, or have a vasectomized partner (confirmed sterile).

   Women with tubal ligation are required to use one non-hormonal contraceptive method.

   Women who are postmenopausal for at least 2 years, and women with total hysterectomy are considered of non-childbearing potential.
10. A positive pregnancy test or breast feeding at screening.
11. Participation in an investigational drug trial within 90 days prior to the first intake of trial medication.
12. Donation of blood or plasma within 60 days preceding the first trial-related blood drawing.
13. Subjects with the following laboratory abnormalities at screening as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events ("DAIDS grading table") and in accordance with the normal ranges of the trial clinical laboratory:

    * serum creatinine grade 1 or greater (≥ 1.1 x upper limit of laboratory normal range [ULN]);
    * lipase or pancreatic amylase grade 1 or greater (≥ 1.1 x ULN);
    * hemoglobin grade 1 or greater (≤ 10.9 g/dL)
    * platelet count grade 1 or greater (≤ 124.999 x 109/L);
    * absolute neutrophil count grade 1 or greater (≤ 1.3 x 109/L);
    * aspartate aminotransferase (AST) or alanine aminotransferase (ALT) grade 1 or greater (≥ 1.25 x ULN);
    * total bilirubin grade 1 or greater (≥ 1.1 x ULN),
    * any other laboratory abnormality of grade 2 or above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Fichtenbaum, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati AIDS Clinical Trials Unit, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the community between September 2008 and March 2009
Pre-assignment Details: 1 subject was excluded based upon elevated triglyceride level prior to randomization
Groups:
- B-Darunavir+Ritonavir Initial Arm: Darunavir+ritonavir x 7 days; Rosuvastatin x 7 days; Combination x 7 days
- A-Rosuvastatin Initial Arm: Rosuvastatin x 7 days; darunavir+ritonavir x 7 days; Combination x 7 days
Period: Overall Study
Arm/Group | B-Darunavir+Ritonavir Initial Arm | A-Rosuvastatin Initial Arm
Started | 8 | 9
Completed | 6 | 6
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B-Darunavir+Ritonavir Initial Arm | A-Rosuvastatin Initial Arm | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (11) | 28 (10) | 28 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Rosuvastatin
Time Frame: 7 days
Population: Analysis of 12 subjects who completed all 3 PK visits
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Rosuvastatin: Rosuvastatin 10 mg daily for 7 days.
- Rosuvastatin-Darunavir-Ritonavir: Rosuvastatin 10 mg daily, Darunavir 600 mg and Ritonavir 100 mg twice daily for 7 days
Arm/Group | Rosuvastatin | Rosuvastatin-Darunavir-Ritonavir
Number analyzed (Participants) | 12 | 12
ng/mL | 6.70 [5.26 to 8.53] | 16.32 [11.78 to 22.61]

2. Primary Outcome: AUC of Rosuvastatin
Time Frame: 7 days
Population: Analysis of 12 subjects who completed all 3 PK visits
Measure: Geometric Mean (90% Confidence Interval); unit: ng*hr/mL
Arm/Group | Rosuvastatin | Rosuvastatin-Darunavir-Ritonavir
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 108.96 [83.85 to 141.6] | 161.24 [124.62 to 208.59]

3. Secondary Outcome: To Investigate the Effect of Rosuvastatin on the Steady State Pharmacokinetics of Darunavir/Ritonavir.
Description: Geometric mean of the Concentration minimum of darunavir and ritonavir in the presence and absence of rosuvastatin.
Time Frame: 45 days
Population: Participants taking all three medications
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Darunavir/Ritonavir+Rosuvastatin: Combination of all three medications
Arm/Group | Darunavir/Ritonavir+Rosuvastatin
Number analyzed (Participants) | 12
ng/mL
  Darunavir Cmin with Rosuvastatin | 2744 [2157 to 3492]
  Darunavir Cmin absent Rosuvastatin | 3235 [2759 to 3794]
  Ritonavir Cmin absent Rousuvastatin | 194 [142 to 266]
  Ritonavir Cmin with Rousuvastatin present | 148 [107 to 204]

4. Secondary Outcome: To Compare the Change in Low-density Lipoprotein (LDL) Cholesterol With Rosuvastatin Therapy Alone, Darunavir/Ritonavir Therapy Alone and With the Co-administration of Rosuvastatin and Darunavir/Ritonavir.
Description: LDL values
Time Frame: 45 days
Population: Individuals taking medications with measurements of LDL
Measure: Median (Inter-Quartile Range); unit: mg/dL
Groups:
- Rosuvastatin Alone: LDL values with rosuvastatin administration
- Darunavir/Ritonavir: LDL values with darunavir/ritonavir administration
- Rosuvastatin+Darunavir/Ritonavir: LDL values with all three medications
Arm/Group | Rosuvastatin Alone | Darunavir/Ritonavir | Rosuvastatin+Darunavir/Ritonavir
Number analyzed (Participants) | 12 | 12 | 12
mg/dL | 85 [55 to 96] | 115 [85 to 148] | 80 [69 to 101]

ADVERSE EVENTS:
Groups:
- Darunavir+Ritonavir: Darunavir 600 mg and ritonavir 100 mg twice daily x 7 days
- Rosuvastatin: Rosuvastatin 10 mg daily x 7 days
- Darunavir, Ritonavir and Rosuvastatin: Darunavir 600 mg and Ritonavir 100 mg twice daily with Rosuvastatin 10 mg daily x 7 days
Arm/Group | Darunavir+Ritonavir | Rosuvastatin | Darunavir, Ritonavir and Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 6/15 | 4/14 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Darunavir+Ritonavir (N=15) | Rosuvastatin (N=14) | Darunavir, Ritonavir and Rosuvastatin (N=12)
Headache (General disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 0 | 0
Skin Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Elevated AST (Hepatobiliary disorders) | 2 | 1 | 1 — Grade I < 2 x ULN
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Elevated CPK (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 — Grade I < 3 x ULN
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 — Grade I: 10-12 gm/dL

LIMITATIONS AND CAVEATS:
No clinical outcome data beyond 7 days is available. Cannot necessarily extrapolate directly to persons with HIV.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No